CLINICAL TRIAL: NCT02036047
Title: The Effectiveness of an Exclusive Cold Snare Polypectomy Snare for the Removal of Diminutive Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Exacto
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Diminutive Colorectal Polyp; Cold Snare Polypectomy; Polypectomy Snare; Complete Resection Rate; Postpolypectomy Bleeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exclusive cold polypectomy snare (Experimental): All colorectal polyps up to 10 mm found except for tiny hyperplastic polyps in the rectum and distal sigmoid colon are removed using an exclusive cold polypectomy snare (Exacto cold snare). The technique is cold snare resection of the polyp without tenting without electrocautery and then suction of the transected polyp into a trap followed by submission to the histological evaluation. The hemostatic clipping is not performed after cold snare polypectomy.
  Interventions: Device: exclusive cold polypectomy snare (Exacto cold snare, product number 00711115)
- regular polypectomy snare (Active Comparator): All colorectal polyps up to 10 mm found except for tiny hyperplastic polyps in the rectum and distal sigmoid colon are removed using a regular polypectomy snare. The technique is cold snare resection of the polyp without tenting without electrocautery and then suction of the transected polyp into a trap followed by submission to the histological evaluation. The hemostatic clipping is not performed after cold snare polypectomy.
  Interventions: Device: Regular polypectomy snare (Snare Master, SD-210U-10)

INTERVENTIONS:
Device: exclusive cold polypectomy snare (Exacto cold snare, product number 00711115)
  Arms: Exclusive cold polypectomy snare
Device: Regular polypectomy snare (Snare Master, SD-210U-10)
  Arms: regular polypectomy snare

SUMMARY:
The use of an exclusive cold polypectomy snare enables a clean cut of diminutive colorectal polyps, resulting in an increase in the complete resection rate and a decrease in the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal polyps up to 10 mm in diameter.

Exclusion Criteria:

* patients are less than 20 years old, pregnant, ASA class III and IV, allergic to propofol used or its components (soybeans or eggs), with poor bowel preparation, and with previous colorectal surgical resection.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Complete resection rate of colorectal polyps | 2 weeks
  The complete resection rate of colorectal polyps based on the pathological examination.

SECONDARY OUTCOMES:
Postpolypectomy bleeding | 2 weeks
  Postpolypectomy bleeding within two weeks after cold snare polypectomy

OTHER OUTCOMES:
The procedure time | 1 day
  The procedure time spent for cold snare polypectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan

REFERENCES:
- [Derived] Horiuchi A, Hosoi K, Kajiyama M, Tanaka N, Sano K, Graham DY. Prospective, randomized comparison of 2 methods of cold snare polypectomy for small colorectal polyps. Gastrointest Endosc. 2015 Oct;82(4):686-92. doi: 10.1016/j.gie.2015.02.012. Epub 2015 Apr 25. PMID 25922251